CLINICAL TRIAL: NCT01063582
Title: Noise of Airplanes a Factor of Risk for the Health of the Heart in Pilots and Crew in Operations of the F16 Airplane
Brief Title: Noise, a Risk for Heart in Airplane Pilots
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Fredesvinda Mendez, Universidad Politecnica de Madrid
Other Study IDs: FMendezV001
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2007-01

CONDITIONS: Pericarditis
Keywords: echocardiogram; electrocardiographic; risk factors; noise
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- fighter pilots f-16: This group is made up of pilots from the F-16 Venezuelan military air force stationed in the Base Vicente Landaeta Gil de Barquisimeto, Lara State.
  Interventions: Other: exposure to occupational noise; Procedure: cardiovascular valuation
- aircraft maintenance personnel f-16: Staff responsible for the preparation of aircraft for the flight and maintenance in the hangar at the airbase Vicente Landaeta Gil de Barquisimeto, Lara. Venezuela
  Interventions: Other: exposure to occupational noise; Procedure: cardiovascular valuation

INTERVENTIONS:
Other: exposure to occupational noise — We performed the measurement of occupational noise exposure through sound level meter and Dosimeter during flight operations of F-16 fighter plane.
  Other Names: occupational noise generated by aircraft miliary
Procedure: cardiovascular valuation — Cardiovascular valuation was performed via electrocardiogram and echocardiographic techniques to correlate the changes observed during exposure to occupational noise
  Other Names: cardiovascular study

SUMMARY:
Study of noise generated by military-type aircraft and equipment maintenance in relation to non-auditory effects that impact with the body of the crew and ground staff can cause cardiac pathologies

Hypothesis of work: The pilots and the technical personnel of maintenance that work before the exhibition of noise generated by planes hunt F-16, or equipments of maintenance of the same ones, present major risk of a cardiac affectation, which demonstrates in changes in the normal pace of the heart, in his function of bomb or in hemodynamic conditions.

DETAILED DESCRIPTION:
The work area military airport is characterized by low frequency noise in sound pressure levels exceeding 100 dB, smashing into the body of pilots and ground staff.

It found variations in the thickness of the pericardium and deviation measures ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* exposure to noise from military aircraft

Exclusion Criteria:

* inactive personal or vacation

Ages: 26 Years to 37 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Group of subjects directly exposed to noise from military aircraft F-16 during its operation and maintenance at the airbase Vicente Landaeta Gil de Barquisimeto. Lara. Venezuela
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2005-02; Primary Completion 2005-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
left ventricular systolic function | one year

SECONDARY OUTCOMES:
electrical disturbance of the heart | 15 days
study of the dimensions of cavities of the heart | 15 days
haemodynamic study of the conditions | 15 days
characterization of ambient sound military aero by Sound Level Meter | 15 days
sensitivity analysis of noise dosimetry | 15 days
subjective perception of noise | 15 days
analysis of clinical background for selection of sample subjects | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fredesvinda M Méndez, MSc, Principal Investigator — Universidad Politecnica de Madrid; Manuel Recuero, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Jarup L, Babisch W, Houthuijs D, Pershagen G, Katsouyanni K, Cadum E, Dudley ML, Savigny P, Seiffert I, Swart W, Breugelmans O, Bluhm G, Selander J, Haralabidis A, Dimakopoulou K, Sourtzi P, Velonakis M, Vigna-Taglianti F; HYENA study team. Hypertension and exposure to noise near airports: the HYENA study. Environ Health Perspect. 2008 Mar;116(3):329-33. doi: 10.1289/ehp.10775. PMID 18335099
- [Background] Andren L, Lindstedt G, Bjorkman M, Borg KO, Hansson L. Effect of noise on blood pressure and 'stress' hormones. Clin Sci (Lond). 1982 Feb;62(2):137-41. doi: 10.1042/cs0620137. PMID 7053913
- [Background] ISO 1990 - International Organization for Standardization. Acoustics-Determination of occupational noise exposure and estimation of noise-induced hearing impairment. ISO 1999:1990 (E) Geneva ISO 1990
- [Background] ISO 1970 -International Organization for Standardization. Acoustics- Guide to international standards on the measurement of airborne acoustical noise and evaluation of its effects on human beings. ISO 2204-70 (E) Geneva ISO 1970.
- [Background] Rosenstock, L. Criteria for a recommended standard: occupational noise exposure. National Institute for Occupational Safety and Health. NIOSH, publication June 1998. 98-126.
- [Result] Tomei F, De Sio S, Tomao E, Anzelmo V, Baccolo TP, Ciarrocca M, Cherubini E, Valentini V, Capozzella A, Rosati MV. Occupational exposure to noise and hypertension in pilots. Int J Environ Health Res. 2005 Apr;15(2):99-106. doi: 10.1080/09603120500061534. PMID 16026021
- [Result] Tomei F, Papaleo B, Baccolo TP, Tomao E, Alfi P, Fantini S. [Chronic noise exposure and the cardiovascular system in aircraft pilots]. Med Lav. 1996 Sep-Oct;87(5):394-410. Italian. PMID 9045028